CLINICAL TRIAL: NCT06661382
Title: Use of Platelet Rich Plasma from Cord Blood Vs Placebo in the Treatment of Vulvar Lichen Sclerosus
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Direzione Ginecologia, Principal Investigator, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FLIPP
Record Dates: First submitted 2023-05-22; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Vulvar Lichen Sclerosus
MeSH Terms: conditions — Vulvar Lichen Sclerosus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Infiltrative treatment with CB-PRP Group (Experimental)
  Interventions: Biological: Infiltrative treatment with CB-PRP
- Placebo infiltrative treatment Group (Placebo Comparator)
  Interventions: Biological: Infiltrative treatment with CB-PRP

INTERVENTIONS:
Biological: Infiltrative treatment with CB-PRP — Injection of CB-PRP or placebo into the vulvar site. Three treatments are planned four weeks apart. Three and six months after the last treatment with CB-PRP/ placebo each participant will be re-evaluated by vulvoscopy and biopsy, and will be given validated questionnaires to assess satisfaction, symptoms, and quality of life, psychological state, and sexual function.

SUMMARY:
Vulvar lichen Sclerosus (VLS) is a cutaneous-mucosal dermatosis that causes in the adult female vulvar itching and burning due to scratching abrasions. Dyspareunia is often associated . The areas most affected are the labia minora, the periclitoral area, the navicular dimple, and the perianal area. The placement of VLS in the context of immune-mediated dermatoses is the basis of the rationale for treatment with high potency topical corticosteroids. However, in some cases, local corticosteroid therapy is not sufficient resulting in a significant impact on the quality of life of the patient. This gives rise to the need to identify new treatments such as regenerative medicine.

The term PRP (Platelet Rich Plasma) is used to describe a blood product generated by a two-step centrifugation process of whole blood of a patient to produce a concentration of platelets in a small volume of plasma. PRP can be produced from autologous, homologous blood or from cord blood (CB-PRP).

Our objective is to evaluate the efficacy of CB-PRP versus placebo in the treatment of VLS.

DETAILED DESCRIPTION:
Lichen Sclerosus (LS) is a cutaneous-mucosal dermatosis characterized by chronic changes in the trophism and maturation of the epithelium and the connective tissue. In females, the vulvar region is affected in about 90% of cases, often constituting the only site involved. In the adult female, the predominant symptoms are vulvar itching and burning due to scratching abrasions. Dyspareunia is an often associated. The clinical course is irregular but progressive and is characterized by periods of relative quiescence alternating with episodes of exacerbation of symptoms. The areas most affected are the labia minora, the periclitoral area, the navicular dimple, and the perianal area. The placement of LS in the context of immune-mediated dermatoses is the basis of the rationale for treatment with high potency topical corticosteroids. However, in some cases, local corticosteroid therapy is not sufficient to achieve adequate compensation of the pathology, and significant changes may set in of the vulvar anatomy resulting in a significant impact on the quality of life of the patient. This gives rise to the need to identify new treatments such a regenerative medicine. The term PRP (Platelet Rich Plasma) is used to describe a blood product blood generated by a two-step centrifugation process of whole blood of a patient to produce a concentration of platelets in a small volume of plasma. In addition to platelets, PRP contains large amounts of chemical mediators that promote angiogenesis, recruitment and proliferation of cells implicated in tissue regeneration and healing. PRP can be produced from autologous, homologous (donor) blood or from cord blood (CB-PRP). The main difference between PRP from peripheral blood (PB-PRP) and that from cord blood concerns the relative amount of growth factors and pro- and anti-inflammatory molecules. CB-PRP has been shown to be advantageous from a therapeutic point of view compared with PB-PRP because it contains higher concentrations of anti-inflammatory molecules. In addition, the use of CB-PRP allows for a final product that is not conditioned by the patient's age and by any associated comorbidities, which may instead compromise the quality of PB-PRP. Finally, the advantages of CB-PRP are related to lower production costs and to the greater ease of product preparation. The preparation process of CB-PRP involves a collection of cord blood following the expulsion of the placenta. The blood is then centrifugated using a two-step process. The final product is then injected on the vulvar surface under vulvoscopic guidance. Treatment with PRP is free of any major side effects. The objective of the following study is to evaluate the efficacy of CB-PRP versus placebo in the treatment of VLS.

ELIGIBILITY:
Inclusion Criteria:

* women with VLS (clinical/histological diagnosis)
* good health conditions
* written informed consent signed and dated by the patient

Exclusion Criteria:

* pregnancy
* coagulopathies, platelet disorders, cardiovascular and/or respiratory diseases
* ongoing major infections
* previous vulvar surgery (e.g., lipostructure and/or previous PRP)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-24 (Actual); Primary Completion 2024-11-24 (Estimated); Study Completion 2024-12-24 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction in treatment group vs placebo group | 3 months
  We expect that women in the cord blood platelets rich plasma group will differ with regard of patient satisfaction through the compilation of the Likert scale: 0 better outcome, 10 worst outcome.

SECONDARY OUTCOMES:
Patient Global Impression of Change in treatment group vs placebo group | 3 months
  We expect that women in the cord blood platelets rich plasma group will differ with regard of impression of global changes using the Patient Global Impression of Change Questionnaire.
  Patient Global Impression of Change is a single item questionnaire measuring the global changes since the start of the study treatment on a 7-point scale (1 better outcome, 7 worst outcome).
Change in symptomatology in treatment group vs placebo group | 3 months
  We expect that women in the cord blood platelets rich plasma group will differ with regard of symptoms (itching, burning, dyspareunia and dysuria) using specific likert scale: 0 no symptoms (better outcome), 10 worst symptoms (worst outcome).
Mucosal trophism in treatment group vs placebo group | 3 months
  We expect that women in the cord blood platelets rich plasma group will differ with regard of objective change of mucosal trophism through vulvoscopy.
Histological biopsy in treatment group vs placebo group | 3 months
  We expect that women in the cord blood platelets rich plasma group will differ with regard of changing of histological byopsy features, trough biopsy.
Sexual activity changes in treatment group vs placebo group | 3 months
  We expect that women in the cord blood platelets rich plasma group will differ with regard of change in sexual life (considering sexual activity and sexual items like desire, orgasm, pain, lubrication and arousal) using Female Sexual Function Index.
Quality of life changes in treatment group vs placebo group | 3 months
  We expect that women in the cord blood platelets rich plasma group will differ with regard quality of life, through Short Form Health Survey (12 items.

CONTACTS AND LOCATIONS:
Overall Officials: veronica Boero, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan, Milan, Italy